CLINICAL TRIAL: NCT03082417
Title: Improving PAIN Control Following FRactures; Towards an Elder-friendly Emergency Department
Brief Title: The PAINFREE Initiative, a Stepped Wedge Cluster Randomized Trial
Acronym: PAINFREE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Research Institute of the McGill University Health Center (Unknown); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Suzanne Morin, Associate Professor, Department of Medicine, McGill University Montreal General Hospital-McGill University Health Centre, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: MP-CUSM-13-054
Record Dates: First submitted 2017-03-06; First posted 2017-03-17 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Elderly; Older Adults; Bone Fracture; Emergency Department; Pain, Acute
Keywords: Bone Fracture; 75 years old; Elderly; Older adults; Pain scale; Pain documentation; Analgesics; Acetaminophen; Opioid; Nonsteroidal anti-inflammatory drugs; Emergency Department
MeSH Terms: conditions — Fractures, Bone; Emergencies; Acute Pain

STUDY DESIGN:
Intervention Model Description: Pragmatic Stepped Wedge Cluster Randomized Trial
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pre-Implementation (No Intervention): Medical records of patients with a fracture visiting the Emergency departments will be reviewed.
  Data will be collected as a baseline prior to the intervention regarding how nurses and physicians working at Emergency Departments manage acute pain in targeted population.
- Implementation (Experimental): In this stepped-wedge trial design, the experimental arm refers to the time period during patients advertising and educational interventions. It consists in:
  Informing patients visiting Emergency department for fracture about Pain Management Nurses and physicians working at the Emergency Departments will receive an educational interventions focused on optimal acute pain management in older adults with fracture.
  Interventions: Other: Implementation
- Post-Implementation (No Intervention): Data will be collected after the intervention regarding how the intervention impacted nurses' and physicians' work in the pain management in older adults with fracture visiting Emergency Departments manage acute pain in older adults.

INTERVENTIONS:
Other: Implementation — The PAINFREE Initiative is a Multifaceted intervention:
  1. Educating and providing point-of-care tools to nurses working at Emergency Department to improve pain management in older adults with fractures
  2. Educating and providing point of care tools to Emergency Departments physicians working at Emergency Department to improve pain management in older adults with fractures
  3. Inform the patients and their family about how to better manage the pain after a fracture
  Arms: Implementation

SUMMARY:
The PAINFREE (Improving PAIN control following FRactures; towards an Elder-friendly Emergency department) Initiative is a patient-centered multifaceted intervention which aims to improve pain management in patients 75 years and older presenting with a fracture at 7 Emergency Department of participating Montreal hospitals:

1. Montreal General Hospital
2. Royal Victoria Hospital
3. Ste Mary's Hospital
4. Hôpital de Verdun
5. Hôpital du Sacré-Coeur de Montréal
6. Jewish General Hospital
7. Lakeshore General Hospital

DETAILED DESCRIPTION:
Using a stepped-wedge cluster randomized trial design, we will implement PAINFREE sequentially in 7 Emergency Departments (EDs) in the greater Montreal area where as each ED site acts as its own control and provides data in both pre- and post-implementation periods. Mixed methods analysis will be used to link quantitative (pain management indicators pre- and post-implementation) to qualitative (feasibility, fidelity and acceptability of implementation) data sets to facilitate data triangulation to evaluate the effects of PAINFREE in real world settings.

PAINFREE Initiative at each site includes 3 phases: pre-implementation, implementation, and post-implementation. The approach is patient-centered and is composed of three complementary components: a patient component, a physician component, and a nursing component.

Each program phases include the following steps:

1. Pre-implementation (2 months):

   1. In all study sites, distribution and analysis of a web-based survey for nurses to document factors that can impact PAINFREE implementation in their environment
   2. Review of medical records of the target population for extraction of selected variables
2. PAINFREE implementation (6 months):

   1. Awareness campaigns will be organized throughout the institution of each study site (posters, brochures, billboards, lanyards)
   2. Profession-specific educational presentations (1 hour) for physicians and nurses, accredited as part of continued professional development programs
   3. Distribution of standardized point-of-care tools to improve pain assessment and documentation (pocket cards, use of validated pain scales), treatment (standardized prescription) and re-assessment
   4. Distribution of educational material and tools targeting pain care literacy (pain scale interpretation, pamphlet) for patients and their families
3. Post-implementation (4 months):

   1. Review of medical records of target population for extraction of selected variables
   2. Distribution of report cards comparing each ED's post- and pre-intervention performance on pain management indicators and comparing their performance to that of other sites
   3. Phone call interviews with patients
   4. Focus group interviews (physicians and nurses)

ELIGIBILITY:
Inclusion Criteria:

* Age 75 years old or older
* Visiting Emergency Departments for a fracture

Exclusion Criteria:

* Having a skull fracture
* Having only fingers or toes fractures

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1375 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
Time to achieve pain score documentation, and/or administration of an analgesic, within 2 hours of triage, in at least 80% of patients. | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)

SECONDARY OUTCOMES:
Documentation of pain score | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
Time to first pain score documentation | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
Effectiveness of analgesia | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
  Patients with pain score ≥7 who have pain score reduced by ≥ 3 points within 1 hour
Type of analgesia used | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
Mean length of stay in Emergency Department | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
Return to the Emergency Department within 7 days after the first Visit with an uncontrolled pain due to the fracture | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)
Evidence of worsening of Patients mental status while in Emergency Department | Pre-implementation (baseline) and at 6 to 8 months (post-implementation)

OTHER OUTCOMES:
Predictors of successful implementation | at 6 to 8 months after the implementation (post-implementation)
  Qualitative Analysis: Nurses and physicians perceptions and behaviors toward pain management in older adults with fracture at Emergency Department
Change from immediate post-implementation time to analgesia administration at 2 months (end of post-implementation period) | 2 months (end of post-implementation period)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Morin, Dr, Principal Investigator — McGill University Hospital Center
Locations (1):
- Department of Internal Medicine, Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided